CLINICAL TRIAL: NCT05536960
Title: Dotatate to Locate Coronary Plaques at High-risk of Myocardial Infarction
Acronym: DOLPHIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, E.S.stroes, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL80263.018.21
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Atheroscleroses, Coronary
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Dotatate PET/CT (Experimental): These patients will undergo a 68Ga-Dotatate PET/CT scan.
  Interventions: Other: 68Ga-Dotatate PET/CT

INTERVENTIONS:
Other: 68Ga-Dotatate PET/CT — One 68Ga-Dotatate PET/CT to determine uptake of tracer in the arterial wall.

SUMMARY:
To assess whether vulnerable coronary plaques have more uptake of 68Ga-Dotatate than non-vulnerable plaques.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and older
* Underwent CCTA imaging within 78 weeks from the screening visit
* Either CAD-RADS 4 or higher or 0/1 on CCTA.
* Able to provide written informed consent

Exclusion Criteria:

* History of chronic kidney disease stage 3b - 5, defined as a CKD-EPI value of < 45 ml/min/1,73m2.
* CVD events/revascularization in history
* Malignant diseases or any clinically significant medical condition that could interfere with the conduct of the study in the opinion of the investigator.
* Chronic or recent (< 1 month) infections and/or clinical signs of acute infection.
* History of auto-immune diseases.
* Standard contra-indications to 68Ga-Dotatate PET, and CT based on physicians experience and current practices.
* Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.
* Elevated liver enzymes (> 2 ULN of liver transaminases), acute liver failure or known liver disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Difference in TBRmax | 1 day
  Difference of target to background ratio (TBR)max in the coronary arteries between groups.

SECONDARY OUTCOMES:
Correlation between TBRmax and FAI. | 1 day
  Correlation of TBRmax with fat attenuation index, a specific CCTA parameter of vascular inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No